CLINICAL TRIAL: NCT02032173
Title: A 24 Month Open-label, Multicenter, Phase IIIb Study of the Efficacy and Safety of Lucentis® (Ranibizumab 0,5mg) in Diabetic Patients With Visual Impairment Due to Macular Edema Evaluating a Spaced Out Follow-up After Intensive Loading Phase
Brief Title: Efficacy and Safety of Lucentis® Use in Patients With Diabetic Macular Edema Evaluating a Spaced Out Follow-up After Intensive Treatment Phase
Acronym: CONSTELLATION
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was prematurely discontinued as it was unethical to continue based on a change in ranibizumab (RFB) marketing authorization.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002DFR11
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Macular Edema; Macular Degeneration; Diabetes
Keywords: Ranibizumab; Diabetic Macular Edema
MeSH Terms: conditions — Macular Edema; Macular Degeneration; Diabetes Mellitus | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranibizumab 0.5mg (Experimental): Intravitreal injection with standard dose of 0.5 mg/0.05mL Pro re nata (PRN)
  Interventions: Drug: Ranibizumab 0.5mg

INTERVENTIONS:
Drug: Ranibizumab 0.5mg — Intravitreal injection with standard dose of 0.5 mg/0.05mL Pro re nata (PRN)

SUMMARY:
The study was designed to assess the efficacy and safety of Lucentis® (ranibizumab 0.5 mg) in diabetic patients presenting with reduced visual acuity due to diabetic macular edema and evaluating spacing out of follow-up after initial intensive treatment phase.

DETAILED DESCRIPTION:
This was a multicenteric, open-label, phase IIIb study, which comprised of 2 groups: the Main Group and the Rescue Group.

Patient's eligibility was assessed during a screening visit (Visit 1) which took place 14 days maximum before treatment initiation (Visit 2 [Day 0]). All patients were initially included in the Main Group and were to receive an initial loading treatment (6 injections during the intensive treatment phase i.e. every month from Day 0 to Month 5, followed by 2 additional injections at Months 8 and 11). Patients were to be followed-up every 3 months for 18 months (spaced-out follow-up period). Their visual acuity was to be checked at each study visit (Months 3, 6, 8, 11, 14, 17, 20, and 23) to assess their response to treatment. Patients who responded to treatment were maintained in the Main Group. Patients who did not meet pre defined criteria were moved to the Rescue Group and treated at the investigator's discretion.

The trial was terminated before any patient reached month 12.

ELIGIBILITY:
Inclusion Criteria:

* Type I or type II diabetes with HbA1c≤10%
* Visual impairment due to a diabetic macular edema
* Stable antidiabetic treatment (since more than 3 months) or hygiene-dietary

Exclusion Criteria:

* Inflammation or infection in one eye
* Women of childbearing potential without an efficient contraception, pregnant or breastfeeding

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-05-19 (Actual); Primary Completion 2015-04-29 (Actual); Study Completion 2015-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- France (8):
  - Novartis Investigative Site, Bobigny, Seine Saint Denis
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 10 centers across France.
Groups:
- Ranibizumab: Intravitreal injection with standard dose of 0.5 mg/0.05mL Pro re nata (PRN)
Period: Overall Study
Arm/Group | Ranibizumab
Started | 31
Included Population - Main Group (Included population with evaluable patients at specific time points) | 31
Rescue Group (Participants who did not meet the pre-defined criteria were moved to Rescue Group) | 1 (1 participant moved to Rescue Group at M6 and trial discontinued before any data was collected.)
Completed | 0
Not Completed | 31
Not completed — Discontinuation due to sponsor decision | 31

BASELINE CHARACTERISTICS:
Arm/Group | Ranibizumab
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (7.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Stable BCVA in the Study Eye at 24 Months Compared With BCVA at 6 Months
Description: Best-Corrected Visual Acuity (BCVA) letters were measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. A positive change from baseline of BCVA indicates improvement. Best value on the scale 100, worst 0. The number of participants with a stable BCVA (BCVA score at 6 months minus BCVA score at 24 months ≤4 letters) were reported.
Time Frame: Month 6 and 24
Population: Included population: No subjects included as analysis required data at month 24 and trial terminated before any subject reached month 12
Arm/Group | Ranibizumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With a Stable BCVA in the Study Eye at 24 Months Compared With BCVA at 11 Months
Description: Best-Corrected Visual Acuity (BCVA) letters were measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. A positive change from baseline of BCVA indicates improvement. Best value on the scale 100, worst 0. The number of participants with a stable BCVA (BCVA score at 11 months minus BCVA score at 24 months ≤4 letters) was calculated as well as its confidence interval at 95%.
Time Frame: Month 11 and 24
Population: as for outcome 1
Arm/Group | Ranibizumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Visual Acuity: Number of Participants Keeping a BCVA Score Gain ≥10 Letters
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. A positive change from baseline of BCVA indicates improvement. Best value on the scale 100, worst 0. The number of participants maintaining ≥10 letters gains in BCVA (compared to the baseline BCVA [Day 0]) value for each visit from Month 3 onwards were reported.
Time Frame: Baseline, Month 3, 6, 8 and 11
Population: Included population with evaluable patients at specific time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab
Number analyzed (Participants) | 21
Participants
  Month 3 | 8
  Month 6: number analyzed (Participants) | 9
  Month 6 | 4
  Month 8: number analyzed (Participants) | 5
  Month 8 | 3
  Month 11: number analyzed (Participants) | 1
  Month 11 | 1

4. Secondary Outcome: Visual Acuity: Number of Participants Keeping a BCVA Score Gain ≥15 Letters
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. A positive change from baseline of BCVA indicates improvement. Best value on the scale 100, worst 0. The number of participants maintaining ≥15 letters gains in BCVA (compared to the baseline BCVA [Day 0]) value for each visit from Month 3 onwards were reported.
Time Frame: Baseline, Months 3, 6, 8 and 11
Population: Included population with evaluable patients at specific time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab
Number analyzed (Participants) | 21
Participants
  Month 3 | 4
  Month 6: number analyzed (Participants) | 9
  Month 6 | 3
  Month 8: number analyzed (Participants) | 5
  Month 8 | 1
  Month 11: number analyzed (Participants) | 1
  Month 11 | 0

5. Secondary Outcome: Visual Acuity: Number of Participants With a BCVA Loss ≥15 Letters at Months 8 and 11 Compared to Month 6 in the Study Eye.
Description: Best-Corrected Visual Acuity (BCVA) letters were measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. A positive change from baseline of BCVA indicates improvement. Best value on the scale 100, worst 0. Number of participants presenting with a ≥15 letter loss in BCVA (compared to the value observed at 6 months) and leading to a treatment change (Rescue Group) for month 8 and 11 were analyzed.
Time Frame: Months 6, 8 and 11
Population: Included population with evaluable patients at specific time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab
Number analyzed (Participants) | 5
Participants
  Month 6 to Month 8 | 0
  Month 6 to Month 11: number analyzed (Participants) | 1
  Month 6 to Month 11 | 0

6. Secondary Outcome: Visual Acuity : Change of BCVA From Baseline in the Study Eye (ETDRS)
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. A positive change from baseline of BCVA indicates improvement. Best value on the scale 100, worst 0. The mean variation in BCVA was compared to the baseline BCVA value [Day 0] over a period of 24 months for patients in the Main Group.
Time Frame: Baseline, months 1, 2, 3, 4, 5, 6, 8 and 11
Population: Included population with evaluable patients at specific time points.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab
Number analyzed (Participants) | 31
Letters
  Month 1 | 5.45 (6.444)
  Month 2 | 5.81 (7.328)
  Month 3: number analyzed (Participants) | 21
  Month 3 | 8.05 (6.704)
  Month 4: number analyzed (Participants) | 18
  Month 4 | 9.94 (5.805)
  Month 5: number analyzed (Participants) | 16
  Month 5 | 9.88 (5.290)
  Month 6: number analyzed (Participants) | 9
  Month 6 | 11.00 (8.485)
  Month 8: number analyzed (Participants) | 5
  Month 8 | 10.40 (5.413)
  Month 11: number analyzed (Participants) | 1
  Month 11 | 10.00 (NA) — standard deviation not calculated for n=1

7. Secondary Outcome: Central Retinal Thickness : Change of Log OCT From Baseline in the Study Eye
Description: Retinal thickness is assessed by optical coherence tomography (OCT) in the study eye. The retina is the light-sensitive part of the eye. OCT is a laser-based, noninvasive, diagnostic system providing high-resolution, three-dimensional images of the retina. A negative mean change from baseline indicates an improvement and a positive mean change from baseline indicates a worsening.The absolute variations of the Central Retinal Thickness (CRT) was measured using a Spectral Domain-Optical Coherence Tomography (SD-OCT) at each visit. Values were calculated as a log OCT (=log[CRT/200]).
Time Frame: Baseline, months 1, 2, 3, 4, 5, 6, 8 and 11
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log[μm/200]
Arm/Group | Ranibizumab
Number analyzed (Participants) | 31
log[μm/200]
  Month 1 | -0.10 (0.117)
  Month 2 | -0.12 (0.122)
  Month 3: number analyzed (Participants) | 21
  Month 3 | -0.13 (0.123)
  Month 4: number analyzed (Participants) | 18
  Month 4 | -0.13 (0.104)
  Month 5: number analyzed (Participants) | 16
  Month 5 | -0.16 (0.096)
  Month 6: number analyzed (Participants) | 10
  Month 6 | -0.15 (0.120)
  Month 8: number analyzed (Participants) | 5
  Month 8 | -0.12 (0.062)
  Month 11: number analyzed (Participants) | 1
  Month 11 | -0.13 (NA) — standard deviation not calculated for n=1

8. Secondary Outcome: Visual Acuity : Change of BCVA From Baseline in the Study Eye (ETDRS) - Rescue Group
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. A positive change from baseline of BCVA indicates improvement. Best value on the scale 100, worst 0. The mean variation in BCVA was compared to the baseline BCVA value [Day 0] over a period of 24 months for patients in the Rescue Group.
Time Frame: Baseline, Months 3, 6, 8 and 11
Population: Included population for subjects entering Rescue Group: No subjects provided evaluable data after switching to the Rescue Group
Arm/Group | Ranibizumab
Number analyzed (Participants) | 0

9. Secondary Outcome: Central Retinal Thickness : Change of Log OCT From Baseline in the Study Eye - Rescue Group
Description: Retinal thickness is assessed by optical coherence tomography (OCT) in the study eye. The retina is the light-sensitive part of the eye. OCT is a laser-based, noninvasive, diagnostic system providing high-resolution, three-dimensional images of the retina. A negative mean change from baseline indicates an improvement and a positive mean change from baseline indicates a worsening.The absolute variations of the Central Retinal Thickness (CRT) measured using a Spectral Domain-Optical Coherence Tomography (SD-OCT) at each visit. Values were calculated as a log OCT (=log[CRT/200]).
Time Frame: Baseline, Months 3, 6, 8 and 11
Population: as for outcome 8
Arm/Group | Ranibizumab
Number analyzed (Participants) | 0

10. Secondary Outcome: Evaluation of the Spaced Out Follow-up on Visual Functions and Quality of Life
Description: The global score obtained on the Visual Function Questionnaire 25 (VFQ 25) was compared from baseline to months 11 and 24 for the Main group and from baseline to months 12 and 24 for the Rescue group.
Time Frame: baseline, months 11, 12 and 24
Population: as for outcome 1
Arm/Group | Ranibizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the patient screening onwards. However, a safety observation period which started from first injection until 4 weeks after discontinuation - up to 11 months.
Arm/Group | Ranibizumab
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 2/31
Other Adverse Events (participants affected / at risk) | 12/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (N=31)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (N=31)
Coronary artery stenosis (Cardiac disorders) | 1
Eye allergy (Both eyes) (Eye disorders) | 1
Halo vision (Study eye) (Eye disorders) | 1
Macular oedema (Contralateral eye) (Eye disorders) | 1
Posterior capsule opacification (Contralateral eye) (Eye disorders) | 1
Vitreous haemorrhage (Study eye) (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Conjunctivitis (Both eyes) (Infections and infestations) | 1
Conjunctivitis viral (Study eye) (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 1
Wound (Injury, poisoning and procedural complications) | 1
Paraesthesia (Nervous system disorders) | 1
Microalbuminuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.